CLINICAL TRIAL: NCT05022836
Title: Should Four-limb Blood Pressures be Used in Infants With High Risk of Congenital Malformation of Aorta?
Brief Title: Four-limb Blood Pressures in Infants With High Risk of Congenital Malformation of Aorta
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yifei WANG, Deputy director of the Neonatology Department, Principal Investigator, Guangdong Provincial People's Hospital
Other Study IDs: Four-limb BPs in CMoA
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Congenital Heart Disease in Children; Coarctation of Aorta; Interrupted Aortic Arch; Hypoplasia of Aorta; Blood Pressure
Keywords: Congenital Heart Disease; Coarctation of Aorta; Interrupted Aortic Arch; Hypoplasia of Aorta; Blood Pressure; screening
MeSH Terms: conditions — Aortic Coarctation; Heart Defects, Congenital | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: four-limb blood pressure measurements — Four-limb blood pressures were measured by certificated nurses at admission.
  Other Names: Echocardiogram or cardiac computed tomography results were used as the gold standard.

SUMMARY:
Pulse oximetry screening (POS) for critical congenital heart diseases (CCHD) could identify 90% of these infants. However, this approach is not designed to detect cardiac defects without hypoxemia, especially congenital malformations of aorta (CMoA). More than 60% of CMoA was late diagnosed.

Infants with CMoA were supposed to present with blood pressure (BP) gradient between four limbs. But a large sample size retrospective study of four-limb BP screening showed a negative result. The possible reason is that this study ran in population with a very low risk of CMoA. Whether four-limb BPs measurement could be used in infants with high risk of congenital malformation of aorta is still to be determined.

The investigators retrospectively collected four-limb BPs, which was prospectively measured, in infants with high risk of CMoA. These data were divided into two groups, the discovery group and the validation group. The best cutoff of four-limb BP gradient was generated by Youden Index. The BP gradients by age were analyzed. Pre-operative hypotension and post-operative hypertension were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the Guangdong Provincial People's Hospital between January 1st, 2013 and December 31st, 2019, who were suspected as having congenital heart disease, were enrolled in the study.

Exclusion Criteria:

* Infants without four-limb blood pressures measurement or without echocardiogram and cardiac computed tomography results were excluded.

Ages: 0 Days to 1 Year | Sex: All
Age Groups: Child
Study Population: Infants admitted to the Guangdong Provincial People's Hospital between January 1st, 2013 and December 31st, 2019, who were suspected as having congenital heart disease, were enrolled in the study. Four-limb BPs in infants of confirmed or suspected CCHD admitted at our hospital were prospectively collected at admission following the Pediatric Department protocol for CCHD infants in which all infants with high risk of CCHD, defined as confirmed or suspected CCHD by clinical teams, were screened by measuring four-limb BPs by certificated nurses. Suspected CCHD was defined as unreasonable low SpO2, cyanosis, murmur, suspected CHD by prenatal ultrasound or postnatal echocardiography at other hospitals, and unexplained poor cardiac output.
Sampling Method: Non-Probability Sample
Enrollment: 1604 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
The cutoff of four-limb BPs gradient to diagnose CMoA | at admission
  ROC curve and Youden Index were used in the discovery group and the validation group to spot the optimal cutoff of BP gradient.

SECONDARY OUTCOMES:
The accuracy of four-limb BPs measurement to predict CMoA | at admission
  The sensitivity, specificity, Youden index, the area under the ROC curve, likelihood ratio for positive test results, likelihood ratio for negative test results, positive predictive value, and negative predictive value were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Yifei Wang, MD, Principal Investigator — Guangdong Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided